CLINICAL TRIAL: NCT00587977
Title: ECG-Gated Multidetector CT of Aortic Distensibility FAMRI
Brief Title: Aortic Distensibility
Acronym: FAMRI
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Joel Garland Fletcher, M.D., Mayo Clinic Rochester, Minnesota
Other Study IDs: 1994-04; 2A3360; FAMRI 2
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Aortic aneurysm repair
- 2: Aortic aneurysm growth
- 3: Aortic aneurysm growth stable.

SUMMARY:
Can software be developed to automatically aid in the measurement of abdominal aortic aneurysms, and is there a way to predict future rupture or growth of abdominal aortic aneurysms.

DETAILED DESCRIPTION:
Hypothesis: ECG-gated multidetector CT and ECG-gated Dual Source CT can be used to create multiple volumetric datasets of the abdominal aorta over the time period of the cardiac cycle, allowing for direct and regional calculations of abdominal aortic distensibility over the entire volume of the abdominal aorta, providing insight into risk of abdominal aortic aneurysm rupture and early large vessel stiffness.

ELIGIBILITY:
Inclusion Criteria:

* AAA must be at least 3 cm to a maximum 4.9cm cross-sectional diameter.
* BMI 31 or less.
* Creatinine results <2.0 and within six months prior to scan.
* US patients must have only normal creatinine (0.9 to 1.4) for one year before study visit.
* Patients who are originally scheduled for US, who are then subsequently rolled in this study, will have only a ultrasound scan as followup after the initial CTA.

Exclusion Criteria:

* Creatinine > 2.0.
* Creatinine <0.9 or >1.4 for those who are scheduled for US.
* Atrial fibrillation or other arrythmia.
* Known AAA greater than 5 cm in size.
* Allergy to contrast dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing imaging of their abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2004-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
In year one, this data will be used to develop pulsatility software and test robustness. | First Year

SECONDARY OUTCOMES:
In year two, the time-resolved CT angiographic datasets from each patient will be analyzed to determine peak AAA pulsatility and peak AAA relative pulsatility (to cross-sectional area within the aneurysm). | Year Two

CONTACTS AND LOCATIONS:
Overall Officials: Joel G. Fletcher, M.D., Principal Investigator — Mayo Clinic - Rochester, Minnesota
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Zhang J, Fletcher JG, Vrtiska TJ, Manduca A, Thompson JL, Raghavan ML, Wentz RJ, McCollough CH. Large-vessel distensibility measurement with electrocardiographically gated multidetector CT: phantom study and initial experience. Radiology. 2007 Oct;245(1):258-66. doi: 10.1148/radiol.2451060530. PMID 17885194
- [Background] Wentz RJ, Manduca A, Fletcher JG, Siddiki HA, Shields RC, Vrtiska TJ, Spencer GC, Primak AN, Zhang J, Nielson TA, McCollough CH, Yu L. SPIE Medical Imaging 2007.: Physiology, Function, and Structure from Medical Images, 2007; 6511:1-9